CLINICAL TRIAL: NCT03039998
Title: Validity of Biological Material Sampling in Patients With Hospital-acquired Pneumonia
Status: Completed | Type: Observational
Sponsor: University Hospital Olomouc (Other)
Collaborators: Palacky University (Other)
Responsible Party: Principal Investigator, Radovan Uvizl, Radovan Uvízl, MD, PhD, University Hospital Olomouc
Other Study IDs: NT14382
Record Dates: First submitted 2016-05-10; First posted 2017-02-01 (Estimated); Last update posted 2017-02-01 (Estimated); Status verified 2017-01

CONDITIONS: Hospital Acquired Pneumonia
MeSH Terms: conditions — Healthcare-Associated Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — endotracheal aspirate, gastric aspirate, oropharyngeal swab, protected specimen brushing
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- HAP Patients: HAP, intubated and mechanically ventilated.

SUMMARY:
The main objective of project is to compare validity of sampling methods performed routinely (bronchial secretion, stomach content, oropharyngeal smear) for determination of etiological agent responsible for hospital-acquired pneumonia (HAP) in critically ill patients to bronchoscopy-assisted protected brush method. Evaluation of the present clinical praxis using bronchial secretion sampling in HAP diagnostics and detection of the most common etiological agents in patients with HAP are other priorities of the project. Aiming to confirm or exclude the diagnosis of HAP, determine the sources and possible routes of bacterial pathogens transmission molecular biology analysis of etiological agents is performed. Finally, percentage of HAP etiological agents resistant to initial empiric antibiotic therapy will be observed.

DETAILED DESCRIPTION:
The main objective of project will be comparing validity of sampling methods performed routinely (bronchial secretion, stomach content, oropharyngeal smear) for determination of etiological agent responsible for hospital-acquired pneumonia (HAP) in critically ill patients to bronchoscopy-assisted protected brush method. Obtained results of different methods will enable to determine if the bronchial secretion sample, stomach content sample or oropharyngeal smear are comparable to precise but technically difficult protected brush. Evaluation of the present clinical praxis using bronchial secretion sampling in HAP diagnostics and detection of the most common etiological agents in patients with HAP will be other priorities of the project. The role of atypical and fungal pathogens in HAP initiation will be discovered as well. Aiming to confirm or exclude the diagnosis of HAP, determine the sources and possible routes of bacterial pathogens transmission molecular biology analysis of etiological agents will be performed. Finally, percentage of HAP etiological agents resistant to initial empiric antibiotic therapy will be observed.

Project fulfills program objectives of molecular-biologic approaches and research support in infectious diseases domain. It will make contribution to faster and more precise HAP diagnosis and adequate antibiotic therapy.

ELIGIBILITY:
Inclusion Criteria:

* clinical signs of HAP
* need for intubation and mechanical ventilation

Exclusion Criteria:

* inability to obtain samples in 24 hours after clinical diagnosis of HAP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patients hospitalized in the Department of Anesthesiology and Intensive Care Medicine, Faculty of Medicine and Dentistry, Palacky University Olomouc and University Hospital Olomouc fulfilling HAP criteria will be enrolled in the study: presence of newly developed or progressive infiltrates on chest radiographs after minimum of 48hours of hospitalization plus at least two other signs of respiratory tract infection: temperature >38 °C, purulent sputum, leukocytosis >10x103/mm3 or leukopenia <4x103/mm3, signs of inflammation on auscultation, cough and/or respiratory insufficiency with oxygenation index (Horowitz) PaO2/ FiO2 ≤300 mm Hg. Clinically ongoing lung inflammation is verified by chest radiograph or CT in the mechanically ventilated patient.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Sensitivity and specificity of diagnostic methods etiological agents HAP. Scale: sensitivity and specificity of each method. | 72 hours
  Obtaining 4 types of agent samples: endotracheal aspirate, gastric aspirate, oropharyngeal swab and protected specimen brushing when clinical signs of HAP arisen and after 72 hours

CONTACTS AND LOCATIONS:
Overall Officials: Tomáš Gabrhelík, MD, PhD, Principal Investigator — University Hospital Olomouc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent JL, Bihari DJ, Suter PM, Bruining HA, White J, Nicolas-Chanoin MH, Wolff M, Spencer RC, Hemmer M. The prevalence of nosocomial infection in intensive care units in Europe. Results of the European Prevalence of Infection in Intensive Care (EPIC) Study. EPIC International Advisory Committee. JAMA. 1995 Aug 23-30;274(8):639-44. PMID 7637145
- [Background] Uvizl R, Hanulik V, Husickova V, Sedlakova MH, Adamus M, Kolar M. Hospital-acquired pneumonia in ICU patients. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2011 Dec;155(4):373-8. doi: 10.5507/bp.2011.067. PMID 22336651
- [Background] American Thoracic Society; Infectious Diseases Society of America. Guidelines for the management of adults with hospital-acquired, ventilator-associated, and healthcare-associated pneumonia. Am J Respir Crit Care Med. 2005 Feb 15;171(4):388-416. doi: 10.1164/rccm.200405-644ST. No abstract available. PMID 15699079
- [Background] Craven DE, Palladino R, McQuillen DP. Healthcare-associated pneumonia in adults: management principles to improve outcomes. Infect Dis Clin North Am. 2004 Dec;18(4):939-62. doi: 10.1016/j.idc.2004.08.001. PMID 15555833
- [Background] Uvizl R, Adamus M, Cerny V, Dusek L, Jarkovsky J, Sramek V, Matejovic M, Stourac P, Kula R, Malaska J, Sevcik P. Patient survival, predictive factors and disease course of severe sepsis in Czech intensive care units: A multicentre, retrospective, observational study. Biomed Pap Med Fac Univ Palacky Olomouc Czech Repub. 2016 Jun;160(2):287-97. doi: 10.5507/bp.2015.052. Epub 2015 Oct 23. PMID 26526190
- [Background] Jones RN. Microbial etiologies of hospital-acquired bacterial pneumonia and ventilator-associated bacterial pneumonia. Clin Infect Dis. 2010 Aug 1;51 Suppl 1:S81-7. doi: 10.1086/653053. PMID 20597676
- [Background] [Pneumonia-causing bacterial pathogens in intensive care patients]. Klin Mikrobiol Infekc Lek. 2011 Aug;17(4):135-40. Czech. PMID 22052100
- [Background] Torres A, Ewig S, Lode H, Carlet J; European HAP working group. Defining, treating and preventing hospital acquired pneumonia: European perspective. Intensive Care Med. 2009 Jan;35(1):9-29. doi: 10.1007/s00134-008-1336-9. Epub 2008 Nov 7. PMID 18989656
- [Background] Kowalczyk W, Rybicki Z, Tomaszewski D, Truszczynski A, Guzek A. [The comparison of different bronchial aspirate culturing methods in patients with ventilator-associated pneumonia (VAP)]. Anestezjol Intens Ter. 2011 Apr-Jun;43(2):74-9. Polish. PMID 22011866
- [Background] Butler KL, Best IM, Oster RA, Katon-Benitez I, Lynn Weaver W, Bumpers HL. Is bilateral protected specimen brush sampling necessary for the accurate diagnosis of ventilator-associated pneumonia? J Trauma. 2004 Aug;57(2):316-22. doi: 10.1097/01.ta.0000088858.22080.cb. PMID 15345979
- [Background] Gerbeaux P, Ledoray V, Boussuges A, Molenat F, Jean P, Sainty JM. Diagnosis of nosocomial pneumonia in mechanically ventilated patients: repeatability of the bronchoalveolar lavage. Am J Respir Crit Care Med. 1998 Jan;157(1):76-80. doi: 10.1164/ajrccm.157.1.9604070. PMID 9445281